CLINICAL TRIAL: NCT01607632
Title: An Open Pilot Study of Loving-Kindness Meditation for PTSD
Brief Title: Loving-kindness Meditation for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Principal Investigator, David Kearney, Staff Physician, Seattle Institute for Biomedical and Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00173
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress; depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- loving-kindness meditation (Experimental)
  Interventions: Behavioral: loving-kindness meditation

INTERVENTIONS:
Behavioral: loving-kindness meditation — A 12-week duration, 90 minute per session loving-kindness meditation course

SUMMARY:
A before and after study of veterans who took part in a 12-week loving-kindness meditation course as an adjunct to their usual care for posttraumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* posttraumatic stress disorder

Exclusion Criteria:

* psychosis
* borderline personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change in PTSD symptoms | baseline, post-intervention, 3-month follow-up
  The PTSD symptom-scale interview was performed
change in depressive symptoms | baseline, post-intervention, 3-month follow-up
  The PROMIS measure for depression was administered

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — VA Puget Sound
Locations (1):
- VA Puget Sound, Seattle, Washington, United States